CLINICAL TRIAL: NCT04592523
Title: Post-Marketing Surveillance (Usage Results Study) of Brigatinib in the Treatment of Adult Patients for Approved Indications in South Korea
Brief Title: A Study of Usage of Brigatinib in the Treatment of Adult Participants for Approved Indications In South Korea
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brigatinib-5005; U1111-1257-0204 (Registry Identifier: WHO)
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Anaplastic Lymphoma Kinase
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants diagnosed with anaplastic lymphoma kinase (ALK)-positive advanced or metastatic non-small cell lung cancer (NSCLC) who initiate treatment for the first time with brigatinib in a routine clinical practical setting will be observed prospectively for up to 24 month-surveillance period.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The purpose of this study is to estimate the proportion of all adverse events (AEs) including serious adverse events (SAEs) occurring with the use of brigatinib among adult participants who have been administered brigatinib as per the approved indications.

DETAILED DESCRIPTION:
This is a prospective observational post-marketing surveillance study of participants with ALK-positive NSCLC who initiate treatment for the first time with brigatinib in a routine clinical practical setting. The study will characterize the safety and effectiveness of brigatinib for its approved indications under real world use.

The study will enroll approximately 257 participants. The data will be prospectively collected, at the centers from routinely scheduled and emergency visits until end of follow up, and recorded into electronic case report forms (e-CRFs). All participants will be assigned to a single observational cohort.

This multi-center study will be conducted in the South Korea. The overall duration of this study is approximately 6 years. Data will be collected over and up to a 24 month-surveillance period (per participant) once enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. With ALK-positive advanced or metastatic NSCLC.
2. Who initiate brigatinib for the first time.

Exclusion Criteria:

1. Treated with brigatinib outside of the locally approved label in Korea.
2. Whom brigatinib is contraindicated as per product label.
3. Participating in other clinical trials of NSCLC treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with ALK-positive advanced or metasatatic NSCLC who initiate treatment for the first time with brigatinib in a routine clinical practical setting will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with AEs and SAEs | Up to 30 days after the end of treatment (up to 24 months)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  ORR will be evaluated by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR is defined as the percentage of participants who achieved a best response of a complete response (CR) or partial response (PR). CR: defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Duration of Response (DOR) | Up to 24 months
  DOR will be evaluated according to RECIST version 1.1. DOR is defined as duration from the point at CR or PR is reached first until the day the recurrence of cancer or disease progression is confirmed. CR: defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. Progressive disease (PD) is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Progression Free Survival (PFS) | From first administration of study drug to the date of disease progression or death due to any cause (up to 24 months)
  PFS will be evaluated by treating physicians according to RECIST version 1.1. PFS is defined as the time from the date of first dose to the date of first documentation of disease progression or date of death from any cause, whichever occurs first. Progressive disease (PD) is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/5f9465aa296beb001e63bfa6??page=1&idFilter=Brigatinib-5005